CLINICAL TRIAL: NCT00198731
Title: Evaluation of the Effects of Community-based Interventions on Maternal Morbidity in the Early Postpartum Period in Rural Bangladesh
Brief Title: Evaluation of the Effects of Community-based Interventions
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Other Study IDs: H.22.04.09.03.D1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Pregnancy
Keywords: maternal health; Bangladesh; care seeking

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Care Seeking for Obstetric Complication — This is a descriptive study of knowledge, practices and outcomes related to maternal morbidity during pregnancy, childbirth and postpartum.

SUMMARY:
Maternal death is a substantial burden in developing countries. In Bangladesh, recent studies have suggested that a large proportion of women giving birth in rural areas experience pregnancy and delivery related complications. This study, which is set in context where home-birth is the norm, provides the opportunity to provide descriptive information on the self-reported prevalence of maternal behaviors and morbidities during pregnancy, delivery and postpartum periods and to quantify the effects of provision of maternal care interventions through trained community health workers on a few selected maternal behaviors and morbidities.

DETAILED DESCRIPTION:
Maternal mortality is a substantial burden in developing countries. The World Health Organization (WHO) estimates that between 500,000 to 600,000 women die from complications related to pregnancy and childbirth each year, with 99% of these deaths occurring in developing countries (WHO/UNICEF/UNFPA, 2000). It is estimated that pregnancy-related causes result in about one-quarter to one-third of the deaths of women in their reproductive years (Koblinsky, 1995). Improving maternal mortality has received recognition at the global level as evidenced by the inclusion of reducing maternal mortality in the Millennium Development Goals (United Nations, 2004).

Among problems experienced by women related to child-bearing, maternal mortality is the "tip of the iceberg". Consideration of the morbidity associated with pregnancy, delivery and the postpartum period is essential in understanding the burden of diseases due to maternal causes. The WHO estimates that up to 300 million women suffer from short- or long-term illnesses related to pregnancy and childbirth (WHO, 1998). In addition, the WHO estimates that in developing countries, death and disability related to maternal morbidity account for 18.5% of the burden of disease among women of reproductive age (WHO, 1998).

In Bangladesh, recent studies have suggested that a large proportion of women giving birth in rural areas experience pregnancy- and delivery- related complications (NIPORT et al, 2001), and more than 80% of the women suffer from a serious postpartum illness (Goodburn et al, 1994; BIRPERHT, 1994). In the baseline survey for the project "Community-Based Interventions to Reduce Neonatal Mortality in Bangladesh" in Sylhet, a total of 75% of women reported at least one maternal complication during pregnancy, delivery and the postpartum.

There is little evidence as to the effect of maternal care interventions on maternal morbidity. Several studies have evaluated the impact of traditional birth attendant (TBA) training on morbidity and referral rates. In a review of 15 studies on the effects of TBA training programs, Ray and Salihu found an improvement in maternal morbidities in two of the three studies reviewed, and an impact on referral rates in six of the seven studies reviewed (Ray & Salihu, 2004). In a meta-analysis conducted by Sibley et al, there was no effect detected between TBA training and recognition of maternal complications, referral for complications or on maternal compliance with referral (Sibley, Sipe, & Koblinsky, 2004).

Maternal morbidity is a substantial burden on the health of women in Bangladesh and throughout developing countries. Further research is needed to more carefully document the community-based incidence of maternal morbidity and to evaluate program impact on maternal morbidity.

The objectives of this study are to provide data on descriptive information on self-reported maternal morbidities for future planning, and to measure the effect of a package of maternal care interventions by comparing differences in care seeking for perceived complications and the unmet obstetric need (based on major obstetric interventions (MOI) for facility-validated absolute maternal indications (AMI) ) among the three arms, and by comparing anemia rates among the three arms.

ELIGIBILITY:
Inclusion Criteria:

* Qualitative research:
* Women who have given birth within six to twelve months in sthe study area who give consent to participate in the study
* Quantitative research:
* Women who have given birth in the past 4-8 weeks in the study area who give consent to participate in study
* Women who have experienced a major obstetric intervention in the 12 months prior to the survey who give consent to participate in the study
* Family members of women who have died due to a maternal cause in the 12 months prior to the survey who give consent to participate in the study
* All women enrolled in the home care arm of the parent study who agree to have their temperature taken postpartum

Exclusion Criteria:

* there are no exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 1506 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Baqui, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- N/A - community-based study, Beanibazar, Zakigang and Kanaighat, Bangladesh